CLINICAL TRIAL: NCT07194213
Title: Prevelance of Hypercalciuria in Children With Steroid Dependent Nephrotic Syndrome in Sohag University Hospital
Brief Title: Prevelance of Hypercalciuria in Children With Steroid Dependent Nephrotic Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Ewees Elsayed, Ahmed ewees, Sohag University
Other Study IDs: Soh-Med--25-7-8MS
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Steroid-Dependent Nephrotic Syndrome; Hypercalciuria; Steroid Dependent Nephrotic Syndrome; Hupercalciurea
Keywords: Children; Pediatrics
MeSH Terms: conditions — Nephrotic Syndrome; Hypercalciuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with steroid dependent nephrotic syndrome: Participants will undergo urine analysis to measure calcium excretion in order to assess the prevalence of hypercalciuria. No experimental treatment will be given.

SUMMARY:
Prevelance of hypercalciurea in children with sterorid dependent nephrotic syndrome

DETAILED DESCRIPTION:
Prevelance of hypercalciurea in steroid dependent nephrotic syndrome

ELIGIBILITY:
Inclusion Criteria:

* - Age between 2 and 16 years.
* Diagnosis of steroid-dependent nephrotic syndrome (according to standard clinical criteria).
* Currently in remission or relapse while on steroid therapy.

Exclusion Criteria:

* - Children with congenital or secondary nephrotic syndrome.
* Presence of other chronic kidney diseases.
* Use of medications that affect calcium metabolism (other than steroids).
* Children with systemic diseases affecting bone or mineral metabolism.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children diagnosed with steroid-dependent nephrotic syndrome who are being followed up at the pediatric nephrology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hypercalciurea | At enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) that underlie the results of the study will be made available upon reasonable request from the principal investigator, after publication of the main results.